CLINICAL TRIAL: NCT07334496
Title: A Randomized, Double-blind, Single-dose, Parallel Comparison Study to Evaluate the Biosimilarity of GLR1044 Injection and Dupilumab Injection (Dupixent®) in Healthy Chinese Adult Male Subjects
Brief Title: A Study to Evaluate the Biosimilarity of GLR1044 Injection and Dupilumab Injection (Dupixent®) in Healthy Adult Male Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GLR1044-AD-101
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Biosimilarity
Keywords: Biosimilarity
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLR1044 injection (Experimental)
  Interventions: Drug: GLR1044 injection
- Dupilumab Injection (Active Comparator)
  Interventions: Drug: Dupilumab Injection

INTERVENTIONS:
Drug: GLR1044 injection — GLR1044 injection 300mg/2.0mL; subcutaneous injection; single dose
  Arms: GLR1044 injection
Drug: Dupilumab Injection — Dupilumab Injection 300mg/2.0mL; subcutaneous injection; single dose
  Arms: Dupilumab Injection

SUMMARY:
This is a randomized, double-blind, single-dose, parallel comparison biosimilarity study conducted in healthy Chinese adult male subjects.

It is planned to enroll 198 male subjects in this study. Eligible subjects will be randomized into 2 dosing groups at 1:1 (GLR1044 group or Dupilumab group), i.e., 99 subjects in each group. Each subject is administered once by subcutaneous injection in the abdomen, during which the subject is required to be hospitalized for 4 days. The safety follow-up will last until D57.

ELIGIBILITY:
Inclusion Criteria:

* 1.Voluntarily sign the informed consent form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and be able to follow the contraindications and restrictions specified in this protocol.

  2. Male subjects aged 18 to 55 years (both inclusive) at the time of signing informed consent forms.

  3. Subjects must agree to use reliable contraception for themselves and their partners during the study and within 6 months after the end of the study (the contraception used should comply with local regulations on the use of contraceptive methods for subjects participating in clinical studies), and not donate sperm for assisted reproductive purposes.

  4. The body mass index (BMI) at screening is 19-26 kg/m2 (both exclusive), and the weight is 55-85 kg (both exclusive).

  5. The results of medical history review, physical examinations, laboratory tests, imaging examinations and ECG at screening/visit 2 (V2) are judged by the investigator to be normal or abnormal but not clinically significant.

No personal history of tuberculosis, no possible previous history of tuberculosis exposure, and no previous and/or current immunomodulatory treatment.

6.No personal history of tuberculosis, no possible previous history of tuberculosis exposure, and no previous and/or current immunomodulatory treatment.

Exclusion Criteria:

* 1.History of drug abuse within 1 year prior to screening, or positive predose drug abuse screening result at Visit 2 (V2); or history of alcohol abuse within 6 months prior to screening, or positive predose alcohol breath test result at V2.

  2. Subjects who smoked > 5 cigarettes/day within 3 months prior to screening or who cannot stop using any tobacco products during the study.

  3. The subject and/or first-degree relatives have a history of venous thromboembolic events or idiopathic venous thromboembolic events before screening.

  4. Presence of sunburn, scar tissue, tattoos, open ulcers or branding at screening that the investigator believes will interfere with the interpretation of adverse skin reactions.

  5. Eye or oral infections at screening, including but not limited to conjunctivitis, blepharitis and oral herpes.

  6. The following medical history with a clear diagnosis in the past or at screening: Subjects with cardiovascular disorders, hematological diseases, respiratory disorders, digestive system diseases, abnormal hepatic function, abnormal renal function, endocrine and metabolic disorders (except for overweight), nervous system disorders or psychiatric disorders, skin and subcutaneous tissue disorders, musculoskeletal system disorders, and immune system disorders, who in the opinion of the investigator should be excluded from the study due to the above-mentioned diseases, or other diseases that may interfere with the interpretation of study results.

  7. The estimated glomerular filtration rate at screening is < 90 mL/min/1.73m2 as calculated using the CKD-EPI equation.

  8. Any malignant tumor suspected or diagnosed prior to screening. 9. Subjects with blood donation or blood loss ≥ 400 mL within 3 months prior to screening, or subjects with bone marrow donation.

  10. Subjects who have undergone major surgery (including but not limited to surgery requiring general anesthesia) or organ transplantation within 3 months prior to screening, or are still in a state of illness, trauma or incomplete recovery from surgery at the time of screening (e.g., significant impairment in daily living or working capacity compared to pre-illness/injury/surgery status), or plan to undergo surgery during the study or within two months after the end of the study.

  11.Subjects with allergic constitution, or a history of allergic diseases such as bronchial asthma, urticaria, and eczema.

  12. Known or suspected intolerance or hypersensitivity to any biological drug and its excipients, or known allergy or clinically significant reaction to murine-derived, chimeric, or humanized proteins in monoclonal antibodies or antibody fragments.

  13. Subjects who tested positive for human immunodeficiency virus (HIV) antigen antibody, treponema pallidum antibody, hepatitis B surface antigen (HBsAg) quantitative assay, hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) antibody at screening.

  14.Use of Dupilumab Injection and other cytokine (including but not limited to tumor necrosis factor, interleukin, etc.) targeted agents before screening, or use of other drugs that may affect the judgment of this study result within 3 months before screening (including but not limited to Janus kinase (JAK) inhibitor, phosphodiesterase-4 inhibitor, Fc receptor antagonists (Rozanolixizumab, Efgartigimod, etc.), any biological drugs and preparations, etc.); or have used any biological agent containing immunoglobulins within 1 year before screening.

  15.Subjects who have participated in any clinical trial of an unmarketed drug or vaccine and received medication within 3 months before screening or within 5 half-lives of the previous investigational medicinal product (whichever is longer), or subjects who plan to be vaccinated during the study period or within 2 months after the end of the study.

  16. Subjects who have used prescription and over-the-counter (OTC) drugs, herbal medicines, traditional Chinese medicines, and Chinese patent medicines without the approval of the investigator within 14 days before administration at Visit 2 (V2).

  17. Those who are investigators or employees of the study site, or family members of the employees or investigators.

  18. The investigator believes that there is any condition that may cause the subject to be unable to complete this study or bring obvious risks to the subject, or other investigators believe that the subject has any condition that makes him/her unsuitable for participating in this study, or the subject may not be able to complete this clinical trial for other reasons.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic indicators:Cmax | Day 1-Day 57
Pharmacokinetic indicators:AUC0-∞. | Day 1-Day 57

SECONDARY OUTCOMES:
Pharmacokinetic indicators: AUC0-t | Day 1-Day 57
Pharmacokinetic indicators: CL | Day 1-Day 57
Pharmacokinetic indicators: λz | Day 1-Day 57
Pharmacokinetic indicators: Tmax | Day 1-Day 57
Pharmacokinetic indicators: t1/2 | Day 1-Day 57
Pharmacokinetic indicators: Vz | Day 1-Day 57
Pharmacokinetic indicators: MRT | Day 1-Day 57
Pharmacokinetic indicators: AUC0-t/AUC0-∞ ratio. | Day 1-Day 57
Safety: Number of treatment-emergent adverse events (TEAEs) | Day 1-Day 57
Safety: Number of treatment-emergent serious adverse events (TESAEs). | Day 1-Day 57
Immunogenicity: Anti-drug antibody (ADA) | Day 1-Day 57
Immunogenicity: neutralizing antibody (NAb) | Day 1-Day 57

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gobroad Hospital, Beijing, Beijing Municipality, China